CLINICAL TRIAL: NCT05503394
Title: A Peer Support Network System Construction for the Primary Caregivers of Children With Biliary Atresia Based on Social Support Theory: A Quasi-experimental Study
Brief Title: A Peer Support Network System Construction for the Primary Caregivers of Children With Biliary Atresia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021390
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Biliary Atresia Congenital Type 3

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer support WeChat platform intervention group (Experimental): Peer support WeChat platform intervention for primary caregivers of children with biliary atresia based on routine care during the postoperative period up to one month postoperatively
  Interventions: Behavioral: Peer support WeChat platform intervention; Behavioral: Routine nursing care group
- Routine nursing care group (Other): Perform routine nursing care for primary caregivers of children with biliary atresia during the postoperative period up to one month postoperatively
  Interventions: Behavioral: Routine nursing care group

INTERVENTIONS:
Behavioral: Peer support WeChat platform intervention — Primary caregivers of children with biliary atresia are selected as the study population and divided into intervention and control groups in chronological order at a children's hospital in Shanghai. Primary caregivers who visit the hospital between August 2022 and October 2022 are assigned to the control group and primary caregivers who visit the hospital between January 2023 and March 2023 are assigned to the intervention group. The intervention group will receive a peer support WeChat platform intervention from the day of surgery to one month postoperatively. The level of negative emotions and caregiver burden will be compared between the two groups after the intervention. The intervention group receives the same routine care as the control group.
  Arms: Peer support WeChat platform intervention group
Behavioral: Routine nursing care group — Provide routine inpatient education and post-discharge follow-up to primary caregivers of biliary atresia.

SUMMARY:
The peer support WeChat platform for primary caregivers of children with biliary atresia can provide social support ,help them adopt positive coping styles to face the disease, and reduce negative emotions and caregiver burden.

DETAILED DESCRIPTION:
The primary caregivers of children with biliary atresia have a heavy psychological burden, but there is a lack of supportive research on this population. Therefore, this study used a web-based peer support platform to intervene in the primary caregivers of children with biliary atresia to reduce the psychological burden of this population.

The study consisted of two parts. First, a literature analysis, semi-structured interviews, and expert validation are used to form a peer support WeChat platform for primary caregivers of children with biliary atresia.

Second, primary caregivers of children with biliary atresia are selected as the study population and divided into intervention and control groups in chronological order at a children's hospital in Shanghai. Primary caregivers who visit the hospital between August 2022 and October 2022 are assigned to the control group and primary caregivers who visit the hospital between January 2023 and March 2023 are assigned to the intervention group. The intervention group receives a peer support WeChat platform intervention on top of usual care from the day of surgery to one postoperative month. The levels of negative emotions and caregiver burden are compared between the two groups after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child was diagnosed with biliary atresia congenital type 3 and required kasai portoenterostomy ;
* Providing primary care for the child;
* Use a smartphone and have access to the internet;
* Normal communication ability;
* Volunteering to participate in the study.

Exclusion Criteria:

* Existing or previous mental illness;
* Presence of severe anxiety (SAS ≥ 70 points) or depressive mood (SDS ≥ 70 points);
* Children with comorbidities other than biliary atresia;
* Refusal to cooperate.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
The depression scores in primary caregivers | At the one month after the surgical kasai portoenterostomy
  At the one month after surgical kasai portoenterostomy, primary caregivers' depression scores will be measured using the self-rating depression scale (SDS) by a specially-assigned person. The SDS has a total of 20 items, and the score ranges from 25 to 100 points. The higher the score and the more severe the depression.

SECONDARY OUTCOMES:
The anxiety scores in primary caregivers | At the one month after the surgical kasai portoenterostomy
  At the one month after surgical kasai portoenterostomy, primary caregivers' anxiety scores will be measured using the self-rating anxiety scale (SAS) by a specially-assigned person. The SAS has a total of 20 items, and the score ranges from 25 to 100 points. The higher the score and the more severe the anxiety .

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No